CLINICAL TRIAL: NCT06380322
Title: Stand Ready: Military Health and Nutrition Examination Study
Brief Title: Military Health and Nutrition Examination Study
Acronym: MHANES
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Claire Berryman, Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-034
Record Dates: First submitted 2024-03-30; First posted 2024-04-23 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Type 2 Diabetes; Dyslipidemias; Cardiovascular Diseases
Keywords: Diet Quality; Healthy Eating Index; Body Composition; Dietary Supplements; Gut Microbiome; Army Combat Fitness Test
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Dyslipidemias; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, urine, and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active-duty Army Service Members: All measures will be collected one time during the study, except for the dietary recall (measured two times) and urine sample for total daily energy expenditure using doubly labeled water method (measured 3 time).

SUMMARY:
The Military Health and Nutrition Examination Study (MHANES) is a Department of Defense funded study conducted by Pennington Biomedical Research Center and the US Army Research Institute of Environmental Medicine. This cross-sectional study will assess, in a large, diverse sample of Army Service Members (n=600), food and supplement intake, cardiovascular health, body composition, biomarkers of nutritional status, measures of health status, injury prevalence, mental wellbeing, gut microbiome composition, and physical performance outcomes. The proposed study is modeled after the National Health and Nutrition Examination Survey (NHANES) and customized for the Army population.

DETAILED DESCRIPTION:
Background: Comprehensive scientific data on dietary intake, nutritional status, cardiometabolic health, and performance of a representative sample of active-duty Soldiers are not available. Collecting such data will allow for assessment of disease prevalence and health status, provide novel descriptive information, and examine relationships between health and nutrition variables that are currently unavailable on the Army active-duty population.

Study Aim: To assess, in a large, diverse sample of Army Service Members, dietary intake, nutritional status, cardiovascular health, body composition, metabolic biomarkers of nutritional state, and other measures of health status.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Army Soldiers ≥ 18 years old
* Willing to have biological samples stored for future use
* Willing to have data linked to the Soldier Performance, Health, and Readiness (SPHERE) database

Exclusion Criteria:

* Soldiers under the age of 18 years
* Soldiers with an inability to understand verbal or written instructions or testing materials in English
* Soldiers relocating or getting out of the Army in the next 30 days
* Pregnant females
* Soldiers currently in Basic Training (BCT) and/or One-Station Unit Training (OSUT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active-duty U.S. Army Soldiers (n=600 completers)
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2024-08-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dietary intake | This study will collect one ASA24® recall at visit 1 and a second follow-up 24-hour recall 3-10 days later
  24-hour dietary recalls will be collected using ASA24® to measure intake of macronutrients (protein, carbohydrate, and fat) and micronutrients (vitamins and minerals).
Dietary quality | This study will collect one ASA24® recall at visit 1 and a second follow-up 24-hour recall 3-10 days later
  24-hour dietary recalls will be collected using ASA24®. Diet quality will be assessed by the healthy eating index (HEI).

SECONDARY OUTCOMES:
Depression | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Depression will be assessed by the Patient Health Questionnaire-9 (PHQ-9).
Anxiety | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Anxiety will be assessed by the General Anxiety Disorder-7 (GAD-7) questionnaire.
Resilience | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Resilience will be assessed by the Connor-Davidson Resilience Scale (CD-RISC).
Posttraumatic stress disorder | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Posttraumatic stress disorder (PTSD) will be assessed by the the Primary Care PTSD Screen for DSM-5 (PC-PTSD-5).
Self-efficacy | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Self-efficacy will be assessed by the Generalized Self-Efficacy Scale (GSE).
Mood | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Mood state will be assessed by the Profile of Mood States 2 (POMS2) questionnaire.
Physical activity | ActiGraphs will be administered 0-7 days after study enrollment and worn continuously for 5-7 days.
  Physical activity will be measured using the ActiGraph wGT3X-BT wearable device.
Physical activity | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Physical activity will be assessed by the Physical Activity and Physical Fitness Questionnaire from NHANES.
Physical performance | Data will be collected one time at visit 1 (within 1-2 weeks of study enrollment).
  Participants will self-report their most recent Army Combat Fitness Test (ACFT) results.
Physical injuries | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  A questionnaire on orthopedic injuries will be administered.
Sleep duration and quality | ActiGraphs will be administered 0-7 days after study enrollment and worn continuously for 5-7 days.
  Sleep duration and quality will be measured using the ActiGraph wGT3X-BT wearable device.
Sleep duration and quality | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Sleep duration and quality will be assessed by using the Pittsburgh Sleep Quality Index (PSQI).
Eating behavior (Satiety) | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Assessed using the Satiety scale derived from the validated Military Eating Behavior Survey (MEBS)
Eating behavior (Fast Eating Rate) | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Assessed using the Fast Eating Rate scale derived from the validated Military Eating Behavior Survey (MEBS)
Eating behavior (Slow Eating Rate) | Questionnaires will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  Assessed using the Slow Eating Rate scale derived from the validated Military Eating Behavior Survey (MEBS)
Blood pressure | Measured one time at visit 1 (within 1-2 weeks of study enrollment).
  Measured after an overnight (at least 10 hour) fast, blood pressure will be measured with an automated cuff.
Anthropometric and body composition measures | Measured one time at visit 1 (within 1-2 weeks of study enrollment).
  Height measured using a stadiometer. Body mass and composition (fat mass, percent fat, fat-free mass, skeletal muscle mass, and body water) using bioelectrical impedance analysis, body image scanning, and neck, waist, and hip circumference measurements. If available, at 1-2 Army bases, dual x-ray absorptiometry (DXA) will be used.
Measures of anemia and iron status, nutrient status, hormone status, stress, cardiometabolic health, and inflammation | Measured one time at visit 1 (within 1-2 weeks of study enrollment).
  Measured in blood
Albumin, iodine, and other biomarkers of health | Measured one time at visit 1 (within 1-2 weeks of study enrollment).
  Measured in urine
Gut microbiome composition | Measured one time at visit 1 (within 1-2 weeks of study enrollment).
  Measured in stool
Prescription and over-the-counter medication and supplement use | The information on current use of medications and dietary supplements will be obtained one time at visit 1 (within 1-2 weeks of study enrollment). ASA24® data will be collected at visit 1 and again 3-10 days later
  Volunteers will be asked the name of each supplement and medication used in the past 30 days and the dose, unit, frequency, route, indication, and start/stop date. An opaque bag will be provided to volunteers to transport supplements to the in-person visit. Dietary supplement use will also be assessed by ASA24® in conjunction with the 24-hour dietary recall.
Resting metabolic rate (RMR) | Measured one time at visit 1 (within 1-2 weeks of study enrollment).
  Measured by indirect calorimetry (MedGem or BodyGem indirect calorimeter).
Heart rate variability (HRV) | Measured one time at visit 1 (within 1-2 weeks of study enrollment).
  Heart rate variations will be continuously recorded for 10 minutes with the Zephyr Bioharness™ (Zephyr Technology Corporation, Annapolis, MD, US).
Genomics | Measured one time at visit 1 (within 1-2 weeks of study enrollment).
  Array-based genotyping using blood samples
Hemoglobin mass and blood volume | Measured one time at visit 1 (within 1-2 weeks of study enrollment).
  Hemoglobin mass (Hbmass) will be determined in a subset of participants using the automated CO-rebreathing method. The method is based on the dilution principle where a small volume of tracer (CO) is administered and the subsequent concentration of carboxyhemoglobin (COHb) in the blood allows for calculation of Hbmass.
Total daily energy expenditure (TDEE) | Measured three times, twice at visit 1 (within 1-2 weeks of study enrollment) and third time at day 7.
  Total daily energy expenditure will be assessed by the Doubly Labeled Water (DLW) method. Prior to dosing, volunteers will provide a urine sample that will be used to measure background isotope enrichment. Urine will be collected at 4.5 h and 7 d after dosing. Isotopic elimination rates will be calculated to get the rate of CO2 production. Energy expenditure will be calculated by multiplying the rate of CO2 production by an assumed food quotient of the diet.
Psychomotor Vigilance Test (PVT) | Test will be administered one time at visit 1 (within 1-2 weeks of study enrollment).
  This is a 5-min test of simple visual reaction time widely used to assess alertness. The test requires volunteers to sustain attention and respond to stimuli presented at random intervals on a computer screen by pressing a button. Parameters recorded include reaction time, premature responses, correct responses, and number of lapses.

CONTACTS AND LOCATIONS:
Overall Officials: Claire E Berryman, PhD, RD, Principal Investigator — Pennington Biomedical Research Center
Locations (3):
- United States (3):
  - Fort Campbell, Fort Campbell, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Fort Johnson, Leesville, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karl JP, Margolis LM, Fallowfield JL, Child RB, Martin NM, McClung JP. Military nutrition research: Contemporary issues, state of the science and future directions. Eur J Sport Sci. 2022 Jan;22(1):87-98. doi: 10.1080/17461391.2021.1930192. Epub 2021 Jun 3. PMID 33980120
- [Background] Nindl BC, Jaffin DP, Dretsch MN, Cheuvront SN, Wesensten NJ, Kent ML, Grunberg NE, Pierce JR, Barry ES, Scott JM, Young AJ, O'Connor FG, Deuster PA. Human Performance Optimization Metrics: Consensus Findings, Gaps, and Recommendations for Future Research. J Strength Cond Res. 2015 Nov;29 Suppl 11:S221-45. doi: 10.1519/JSC.0000000000001114. PMID 26506192
- [Background] Rittenhouse M, Scott J, Deuster P. Healthy Eating Index and Nutrition Biomarkers among Army Soldiers and Civilian Control Group Indicate an Intervention Is Necessary to Raise Omega-3 Index and Vitamin D and Improve Diet Quality. Nutrients. 2020 Dec 31;13(1):122. doi: 10.3390/nu13010122. PMID 33396252
- [Background] Eilerman PA, Herzog CM, Luce BK, Chao SY, Walker SM, Zarzabal LA, Carnahan DH. A comparison of obesity prevalence: military health system and United States populations, 2009-2012. Mil Med. 2014 May;179(5):462-70. doi: 10.7205/MILMED-D-13-00430. PMID 24806489
- [Background] Clutter CA, Beckman DJ, Wardian JL, Rittel AG, True MW. Are We Missing an Opportunity? Prediabetes in the U.S. Military. Mil Med. 2024 Jan 23;189(1-2):326-331. doi: 10.1093/milmed/usac197. PMID 35786769
- [Background] Chao SY, Zarzabal LA, Walker SM, Herzog CM, Eilerman PA, Luce BK, Carnahan DH. Estimating diabetes prevalence in the Military Health System population from 2006 to 2010. Mil Med. 2013 Sep;178(9):986-93. doi: 10.7205/MILMED-D-13-00147. PMID 24005548
- [Background] Herzog CM, Chao SY, Eilerman PA, Luce BK, Carnahan DH. Metabolic syndrome in the Military Health System based on electronic health data, 2009-2012. Mil Med. 2015 Jan;180(1):83-90. doi: 10.7205/MILMED-D-14-00039. PMID 25562862
- [Background] Shrestha A, Ho TE, Vie LL, Labarthe DR, Scheier LM, Lester PB, Seligman MEP. Comparison of Cardiovascular Health Between US Army and Civilians. J Am Heart Assoc. 2019 Jun 18;8(12):e009056. doi: 10.1161/JAHA.118.009056. Epub 2019 Jun 5. PMID 31164033
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Prins A, Bovin MJ, Smolenski DJ, Marx BP, Kimerling R, Jenkins-Guarnieri MA, Kaloupek DG, Schnurr PP, Kaiser AP, Leyva YE, Tiet QQ. The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5): Development and Evaluation Within a Veteran Primary Care Sample. J Gen Intern Med. 2016 Oct;31(10):1206-11. doi: 10.1007/s11606-016-3703-5. Epub 2016 May 11. PMID 27170304
- [Background] Schwarzer, R. and Jerusalem, M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON.
- [Background] McNair DM, Lorr M, Droppleman LF. Profile of Mood States Manual. San Diego, CA: Educational and Industrial Testing Service. 1971.
- [Background] US Department of the Army. (2017) Nutrition and Menu Standards for Human Performance Optimization. Army Regulation 40-25.
- [Background] Knapik JJ, Reynolds KL, Hoedebecke KL. Stress Fractures: Etiology, Epidemiology, Diagnosis, Treatment, and Prevention. J Spec Oper Med. 2017 Summer;17(2):120-130. doi: 10.55460/SPMB-1E6L. PMID 28599045
- [Background] Farina EK, Thompson LA, Knapik JJ, Pasiakos SM, McClung JP, Lieberman HR. Physical performance, demographic, psychological, and physiological predictors of success in the U.S. Army Special Forces Assessment and Selection course. Physiol Behav. 2019 Oct 15;210:112647. doi: 10.1016/j.physbeh.2019.112647. Epub 2019 Aug 8. PMID 31401079
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cole RE, Jayne JM, O'Connor K, McGraw SM, Beyl R, DiChiara AJ, Karl JP. Development and Validation of the Military Eating Behavior Survey. J Nutr Educ Behav. 2021 Sep;53(9):798-810. doi: 10.1016/j.jneb.2021.04.467. Epub 2021 Jun 30. PMID 34215517
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Gibson AL, Holmes JC, Desautels RL, Edmonds LB, Nuudi L. Ability of new octapolar bioimpedance spectroscopy analyzers to predict 4-component-model percentage body fat in Hispanic, black, and white adults. Am J Clin Nutr. 2008 Feb;87(2):332-8. doi: 10.1093/ajcn/87.2.332. PMID 18258622
- [Background] Ling CH, de Craen AJ, Slagboom PE, Gunn DA, Stokkel MP, Westendorp RG, Maier AB. Accuracy of direct segmental multi-frequency bioimpedance analysis in the assessment of total body and segmental body composition in middle-aged adult population. Clin Nutr. 2011 Oct;30(5):610-5. doi: 10.1016/j.clnu.2011.04.001. Epub 2011 May 8. PMID 21555168
- [Background] WEIR JB. New methods for calculating metabolic rate with special reference to protein metabolism. J Physiol. 1949 Aug;109(1-2):1-9. doi: 10.1113/jphysiol.1949.sp004363. No abstract available. PMID 15394301
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Background] Knapik JJ, Farina EK, Fulgoni VL, Lieberman HR. Clinically diagnosed iron and iodine deficiencies and disorders in the entire population of US military service members from 1997 to 2015. Public Health Nutr. 2021 Aug;24(11):3187-3195. doi: 10.1017/S1368980021000495. Epub 2021 Feb 5. PMID 33541462
- [Background] Knapik JJ, Farina EK, Fulgoni VL 3rd, Lieberman HR. Clinically-diagnosed vitamin deficiencies and disorders in the entire United States military population, 1997-2015. Nutr J. 2021 Jun 15;20(1):55. doi: 10.1186/s12937-021-00708-2. PMID 34130698
- [Background] Beal SL. Sample size determination for confidence intervals on the population mean and on the difference between two population means. Biometrics. 1989 Sep;45(3):969-77. PMID 2790131
- [Background] Lenth RV. Some Practical Guidelines for Effective Sample Size Determination. American Statistician. 2001;55:187-93.